CLINICAL TRIAL: NCT05811299
Title: Effects of Abdominal Exercises With and Without Kinesio Taping on Abdominal Strength and Quality of Life in Females With Diastasis Recti.
Brief Title: Effects of Abdominal Exercises and Kinesio Taping on Abdominal Strength in Females With Diastasis Recti.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0503
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Diastasis Recti; Kinesio Taping
Keywords: Childbirth; Isometric Contractions; Kinesio Tape; Postpartum Women; Rectus Abdominus.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Exercises and KT intervention (Experimental): (Group A ) will receive kinesio taping with abdominal exercises. 8 sessions for 4 weeks and 2 session will be given in a week.
  Interventions: Other: Kinesio taping; Other: Abominal exercises
- Abdominal exercises (Active Comparator): (Group B) will receive abdominal exercises 8 sessions for 4 weeks and 2 session will be given in a week.
  Interventions: Other: Abominal exercises

INTERVENTIONS:
Other: Kinesio taping — Total of 8 sessions for 4 weeks 2 sessions in a week.
  Arms: Abdominal Exercises and KT intervention
Other: Abominal exercises — Total of 8 sessions for 4 weeks 2 sessions in a week.

SUMMARY:
Diastasis recti is an increase in the gap between the rectus abdominis muscles at the midline caused by anterior abdominal wall weakening. The aim of this study is to evaluate the effects of abdominal exercises with and without Kinesio taping on abdominal strength of females with diastasis recti for their better quality of life. This study will be randomized controlled trial .Subjects with diastasis recti meeting the predetermined inclusion and exclusion criteria will be requested to participate in the study via informed consent. Non probability convenient sampling technique will be used. 46 participants will be randomly allocated to either Group A or Group B .Group A will be treated with Kinesio Taping applied in a criss -cross design for consecutive 3 days with 1 day gap after taping will do abdominal exercises.Group B will be treated with above mentioned abdominal exercises for 1 month. Pre and post assessment of diastasis recti and abdominal strength will be done using caliper method and manual muscle test and quality of life will be assessed by MAPP-QOL questionnaire.Jinnah Hospital will be the setting and SPSS software will be used.

DETAILED DESCRIPTION:
Diastasis recti is an increase in the gap between the rectus abdominis muscles at the midline caused by anterior abdominal wall weakening. Diastasis recti abdominis is most common in the female population during pregnancy and after childbirth. The abdominals are stretched as your uterus expands during pregnancy, and the linea alba thins and pulls apart causes the rectus abdominis muscles to split during pregnancy. The aim of this study is to evaluate the effects of abdominal exercises with and without Kinesio taping on abdominal strength of females with diastasis recti for their better quality of life.

This study will be randomized controlled trial .Subjects with diastasis recti meeting the predetermined inclusion and exclusion criteria will be requested to participate in the study via informed consent. Non probability convenient sampling technique will be used. 46 participants will be randomly allocated to either Group A or Group B via lottery method.Subjects in Group A will be treated with Kinesio Taping applied in a criss -cross design for consecutive 3 days with 1 day gap after taping will do abdominal exercises which consists of abdominal crunch exercise ,Curl up,abdominal isometric contractions ,posterior pelvic tilt ,bridging. perform these exercises twice a week for 10 repititions for 1 month . Group B will be treated with above mentioned abdominal exercises for 1 month. Pre and post assessment of diastasis recti and abdominal strength will be done using caliper method and manual muscle test and quality of life will be assessed by MAPP-QOL questionnaire. Data will be collected from Jinnah Hospital Lahore.The data collected will be analyzed using SPSS 25.

ELIGIBILITY:
Inclusion Criteria

* Post natal till 6 months
* Rectus abdominis diastasis > 2.7 cm at umbilicus
* Age 18 to 40

Exclusion Criteria:

* Pregnant female
* Hernia
* Females with physical and mental illness
* Females with any other medical condition like cardiorespiratory diseases
* History of malignancy
* Urogynecologic disorders
* Females suffering from other gynecological issues such as endometriosis
* Polycystic ovaries syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with diastasis recti.
Enrollment: 38 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Caliper Method | 4 weeks
  Rectus abdominis diastasis will be measured during the postpartum period with a high degree of reliability when a dial callper is used.
MMT | 4weeks
  Manual muscle testing (MMT) based on a grading system of 0 to 5.To check the abdminal strength
MAPP QOL | 4 weeks
  The Maternal Postpartum Quality of Life (MAPP-QOL) instrument consisted of 41 item to check quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital,Gynae department, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gursen C, Inanoglu D, Kaya S, Akbayrak T, Baltaci G. Effects of exercise and Kinesio taping on abdominal recovery in women with cesarean section: a pilot randomized controlled trial. Arch Gynecol Obstet. 2016 Mar;293(3):557-65. doi: 10.1007/s00404-015-3862-3. Epub 2015 Sep 2. PMID 26329802
- [Background] Gluppe SB, Engh ME, Bo K. Immediate Effect of Abdominal and Pelvic Floor Muscle Exercises on Interrecti Distance in Women With Diastasis Recti Abdominis Who Were Parous. Phys Ther. 2020 Aug 12;100(8):1372-1383. doi: 10.1093/ptj/pzaa070. PMID 32302393
- [Background] Radhakrishnan M, Ramamurthy K. Efficacy and Challenges in the Treatment of Diastasis Recti Abdominis-A Scoping Review on the Current Trends and Future Perspectives. Diagnostics (Basel). 2022 Aug 24;12(9):2044. doi: 10.3390/diagnostics12092044. PMID 36140446
- [Background] Boxer S, Jones S. Intra-rater reliability of rectus abdominis diastasis measurement using dial calipers. Aust J Physiother. 1997;43(2):109-114. doi: 10.1016/s0004-9514(14)60405-0. PMID 11676678